CLINICAL TRIAL: NCT06100354
Title: Study of Patient Preferences in Relation to the Fitting of a Personalized and Connected Joint Prosthesis.
Acronym: FKprefPat
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC22.0233 - FKprefPat
Record Dates: First submitted 2023-01-19; First posted 2023-10-25 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2023-10

CONDITIONS: Prosthesis User; Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preference study: Patients answering the questionnaire with choice sets
  Interventions: Other: Answering preference

INTERVENTIONS:
Other: Answering preference — Patients will answer a questionnaire with two possible choices describing several scenario of used of customized and connected prosthesis

SUMMARY:
The goal of this observational study is to learn about patients' preference toward the use of customized and connected prosthesis. The main questions it aims to answer are:

* What is the acceptability of new customization and connectivity technologies by patients?
* Are they all at the same level of acceptability?

Participants will have to answer to a questionnaire of choice.

ELIGIBILITY:
Inclusion Criteria:

* More than 18
* Non opposition expressed
* Should have a hip, knee or shoulder joint replacement

Exclusion Criteria:

* Opposition expressed
* Having already a hip, knee or shoulder joint prosthesis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population is the population that comes for consultation and needs a hip, knee or shoulder replacement.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2025-06-12 (Estimated)

PRIMARY OUTCOMES:
Gathering preferences for a customized and connected prosthesis by Discrete choice analysis, and with a questionnaire called "Discrete Choice Experiment", based on RUT (Random Utility Theory). | 6 month
  Patient will choose one scenario between the two proposed in the eight choice sets. Then, based on RUT (Random Utility Theory), a conditionnal logit and Mixed logit will be used to calculate the beta coefficiants of the attributes that allow to measure the prefered choice relating to the technology tested

SECONDARY OUTCOMES:
Measuring the ease of use of new technologies through ATI (Affinity for Technology Interaction) scale | 6 month
  Several question about the use of technologies by patients in their daily life are asked.
  Scale ranges from 1-2 (very low affinity) to 5-6 (very high affinity).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stindel, PhD, Study Director — Centre Hospitalo Universitaire de Brest
Locations (1):
- Centre Hospitalo Universitaire de Brest, Brest, Brittany Region, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.